CLINICAL TRIAL: NCT05893524
Title: Uppsala-Dalarna Dementia and Gait Project
Acronym: UDDGait™
Status: Recruiting | Type: Observational
Sponsor: Dalarna University (Other)
Collaborators: Uppsala University (Other); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Prof. Anna Cristina Åberg, Professor, Dalarna University
Other Study IDs: HDA2021-00022; PUBCARE2016_122 (Other: Uppsala University, Sweden)
Record Dates: First submitted 2023-05-12; First posted 2023-06-08 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Dementia, Mixed; Dementia Senile; Dementia of Alzheimer Type; Mild Cognitive Impairment; Subjective Cognitive Impairment
Keywords: Timed Up-and-Go, TUG; TUG dual-task; Cognitive tests; Dementia; Mild Cognitive Impairment; Subjective Cognitive Impairment; Alzheimer's disease; Step parameters; Video recorded tests
MeSH Terms: conditions — Dementia; Mixed Dementias; Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients undergoing memory assessments: Patients undergoing memory assessments at two specialist memory clinics (Uppsala University Hospital in Uppsala and Falu Hospital in Falun). This group includes patients with dementia, mild cognitive impairment and subjective cognitive impairment.
  Interventions: Diagnostic Test: Timed Up-and-Go (TUG single-task); Diagnostic Test: Timed Up-and-Go dual-task (TUGdt); Diagnostic Test: Clinical functional assessment
- Cognitively unimpaired community dwelling people: Age matched cognitively unimpaired community dwelling people recruited via advertisements.
  Interventions: Diagnostic Test: Timed Up-and-Go (TUG single-task); Diagnostic Test: Timed Up-and-Go dual-task (TUGdt); Diagnostic Test: Clinical functional assessment
- Cognitively unimpaired community dwelling people recruited for test-retest reliability analysis: Cognitively unimpaired individuals who agreed to participate in a retesting session.
  Interventions: Diagnostic Test: Timed Up-and-Go (TUG single-task); Diagnostic Test: Timed Up-and-Go dual-task (TUGdt); Diagnostic Test: Clinical functional assessment
- Persons with cognitive impairment recruited for test-retest reliability analysis: Patients undergoing memory assessment at Uppsala University Hospital who agreed to participate in a retesting session and community dwelling older persons with self-reported subjective or mild cognitive impairment. This group includes patients with dementia, mild cognitive impairment and subjective cognitive impairment.
  Interventions: Diagnostic Test: Timed Up-and-Go (TUG single-task); Diagnostic Test: Timed Up-and-Go dual-task (TUGdt); Diagnostic Test: Clinical functional assessment

INTERVENTIONS:
Diagnostic Test: Timed Up-and-Go (TUG single-task) — The TUG test is a well-established clinical test of one mobility sequence: rising from an armchair, walking straight ahead, passing a line marked on the floor, turning around, walking back, and sitting down again.
Diagnostic Test: Timed Up-and-Go dual-task (TUGdt) — Two dual-task tests including TUG (TUGdt) were carried out: TUGdt naming animals and TUGdt months backwards. The outcomes registered were: time scores for TUG single-task and both TUGdt tests, TUGdt costs (relative time difference between TUG single-task and TUGdt), number of different animals named, number of months recited in correct order, number of animals per 10 s, and number of months per 10 s.
Diagnostic Test: Clinical functional assessment — The diagnostic procedure was part of the clinical routine for patients undergoing memory assessment and involved a geriatrician's careful evaluation of the patient's history and cognitive testing including Mini-Mental State Examination (MMSE), Clock Drawing Test, Verbal Fluency Test, and Trail Making Test A and B. In addition, all participants carried out short versions of the Geriatric Depression Scale and the General Motor Function Assessment Scale, as well as static balance according to the Bohannon Method, and hand grip strength using a dynamometer.

SUMMARY:
UDDGait™ is a multidisciplinary research project with the overreaching goal of providing an aid for early identification of cognitive impairment and risk of dementia development, thereby providing a basis for adequate symptom relieving and health promoting interventions.

A new concept is investigated for this purpose: a "dual-task-test", which implies the combination of a well-established mobility test (Timed Up-and-Go, TUG) with a simultaneous verbal task (i.e. TUG dual-task, TUGdt). This type of test has been judged as a potential aid for early identification of dementia disease. More research is needed to further examine the test's validity, reliability and predictive capacity.

The overall aim is to investigate if TUGdt is useful as an aid for prediction of dementia disease. To ensure the results, the aim is also to evaluate the test's measurement properties and to generate normative reference values of healthy control persons.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing memory assessment at at Uppsala University Hospital, Sweden
* Patients undergoing memory assessment at at Falu Hospital, Sweden
* Cognitively unimpaired individuals with a Mini Mental State Examination (MMSE) score of > 26

Exclusion Criteria:

* Inability to walk three meters back and forth
* Inability to rise from a sitting position
* Indoor use of a walking aid
* Current or recent hospitalization (within the last 2 weeks)
* Need of an interpreter to communicate in Swedish

Ages: 37 Years to 94 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients have been consecutively included when undergoing memory assessment at two specialist clinics in Sweden during the study recruitment period (April 2015 to February 2017 at Uppsala University Hospital and June 2015 to June 2016 at Falu Hospital).
  Age matched cognitively unimpaired community dwelling individuals without cognitive impairment were recruited through advertisements and flyers (May 2017 to March 2019 in Uppsala).
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2015-04-09 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Conversion to dementia | Upp to 10 years
  Diagnostic information for follow-ups and eventual dates of death, all participants' medical records will be reviewed by an experienced geriatrician. Participants will be classiﬁed as having "converted" after receiving a dementia diagnosis, and as "not converted" when a diagnosis of Subjective or Mild cognitive impairment had been conﬁrmed after baseline, or when a reversion to normal cognition had been stated.
  TUG and TUGdt parameters and composite indices will be examined for association with dementia incidence through Cox regression models with and without adjustment for possible confounding variables such as age, gender, and education. Possible occurrence of gender differences in associations between TUG parameters and dementia incidence will be examined. Optimal cut-off values for predictive TUG parameters (including composite indices) will be estimated. Also, sensitivity, specificity, c-statistics, and Youden's J index will be estimated.

SECONDARY OUTCOMES:
Level of cognitive functioning | Upp to 10 years
  Similarly to TUG and TUGdt parameters, association between different cognitive test results and dementia incidence through Cox regression models with and without adjustment for possible confounding variables such as age, gender, and education will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Cristina Åberg, PhD, Principal Investigator — Dalarna University
Locations (2):
- Sweden (2):
  - Dalarna University, Falun, Dalarna County
  - Uppsala University, Uppsala, Uppsala County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahman HB, Giedraitis V, Cedervall Y, Lennhed B, Berglund L, McKee K, Kilander L, Rosendahl E, Ingelsson M, Aberg AC. Dual-Task Performance and Neurodegeneration: Correlations Between Timed Up-and-Go Dual-Task Test Outcomes and Alzheimer's Disease Cerebrospinal Fluid Biomarkers. J Alzheimers Dis. 2019;71(s1):S75-S83. doi: 10.3233/JAD-181265. PMID 31104024
- [Background] Cedervall Y, Stenberg AM, Ahman HB, Giedraitis V, Tinmark F, Berglund L, Halvorsen K, Ingelsson M, Rosendahl E, Aberg AC. Timed Up-and-Go Dual-Task Testing in the Assessment of Cognitive Function: A Mixed Methods Observational Study for Development of the UDDGait Protocol. Int J Environ Res Public Health. 2020 Mar 5;17(5):1715. doi: 10.3390/ijerph17051715. PMID 32150995
- [Result] Ahman HB, Cedervall Y, Kilander L, Giedraitis V, Berglund L, McKee KJ, Rosendahl E, Ingelsson M, Aberg AC. Dual-task tests discriminate between dementia, mild cognitive impairment, subjective cognitive impairment, and healthy controls - a cross-sectional cohort study. BMC Geriatr. 2020 Jul 29;20(1):258. doi: 10.1186/s12877-020-01645-1. PMID 32727472
- [Result] B Ahman H, Berglund L, Cedervall Y, Kilander L, Giedraitis V, J McKee K, Ingelsson M, Rosendahl E, Aberg AC. Dual-Task Tests Predict Conversion to Dementia-A Prospective Memory-Clinic-Based Cohort Study. Int J Environ Res Public Health. 2020 Nov 3;17(21):8129. doi: 10.3390/ijerph17218129. PMID 33153203
- [Derived] Lofgren N, Giedraitis V, Halvorsen K, Rosendahl E, Aberg AC. The Timed Up and Go dual-task test's cognitive and motor outcomes show promising test-retest reliability in older adults with perceived memory impairment. Front Aging. 2026 Jan 8;6:1715756. doi: 10.3389/fragi.2025.1715756. eCollection 2025. PMID 41585362
- [Derived] Lofgren N, Berglund L, Giedraitis V, Rosendahl E, Aberg AC. Can Turn Duration and Step Parameters During the Timed Up and Go Test With and Without a Dual-Task Discriminate Between Individuals With Different Cognitive Abilities? An Explorative Study. Assessment. 2026 Jan 22:10731911251410337. doi: 10.1177/10731911251410337. Online ahead of print. PMID 41572419
- [Derived] Lofgren N, Berglund L, Giedraitis V, Halvorsen K, Rosendahl E, McKee KJ, Aberg AC. Extracted step parameters during the timed up and go test discriminate between groups with different levels of cognitive ability-a cross-sectional study. BMC Geriatr. 2025 Mar 17;25(1):182. doi: 10.1186/s12877-025-05828-6. PMID 40097949
- [Derived] Aberg AC, Petersson JR, Giedraitis V, McKee KJ, Rosendahl E, Halvorsen K, Berglund L. Prediction of conversion to dementia disorders based on timed up and go dual-task test verbal and motor outcomes: a five-year prospective memory-clinic-based study. BMC Geriatr. 2023 Sep 2;23(1):535. doi: 10.1186/s12877-023-04262-w. PMID 37660032
- See also: Project website — https://www.du.se/en/about-du/organisation/subjects/medicinsk-vetenskap/uddgait-uppsala-dalarna-dementia-and-gait-project/

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT05893524/SAP_000.pdf